CLINICAL TRIAL: NCT01591382
Title: Hydromorphone PCA or Hydromorphone PCA With Ketamine for Acute Postoperative Pain Relief in Opioid-Dependent Chronic Pain Patients
Brief Title: Efficacy Study of Ketamine for Postoperative Pain in Opioid Dependent Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Srdjan Nedeljkovic, Staff, Pain Management Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008P001126
Record Dates: First submitted 2012-05-01; First posted 2012-05-04 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Pain
Keywords: Ketamine; Postoperative pain; Opioid dependent patients; Acute pain control
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Participants received postoperative hydromorphone patient-controlled analgesia (PCA) and continuous ketamine (0.2 mg/kg/hour). Ketamine is being compared to the use of placebo, in addition to intravenous opioids, for postop pain control in opioid dependent patients who undergo major surgery.
  Interventions: Drug: Ketamine; Drug: Hydromorphone PCA
- Placebo (Placebo Comparator): Participants received postoperative hydromorphone PCA and continuous ketamine-matching placebo (infusion of saline).
  Interventions: Drug: Placebo; Drug: Hydromorphone PCA

INTERVENTIONS:
Drug: Ketamine — Intravenous (IV) ketamine 0.2 mg/kg/hr for 24-48 hours postoperatively.
  Arms: Ketamine
Drug: Placebo — Patients who received ketamine-matching placebo were given saline infusions
  Arms: Placebo
Drug: Hydromorphone PCA — Intravenous hydromorphone PCA

SUMMARY:
Patients who are dependent on opioids often have poor pain relief after major surgery. This study tests the hypothesis that adding intravenous ketamine to a postoperative regimen of intravenous opioids for postoperative pain will improve pain relief in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain > 6 months
* Long term use of opioids
* Major surgery

Exclusion Criteria:

* Use of regional anesthetic techniques
* No need for intravenous (IV) patient controlled analgesia (PCA) after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan S Nedeljkovic, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Hydromorphone PCA and ketamine intravenous (IV) infusion 0.2 mg/kg/hr for 24-48 hours postoperatively.
- Placebo: Hydromorphone PCA and placebo-matching ketamine intravenous (IV) infusion 0.2 mg/kg/hr for 24-48 hours postoperatively.
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 32 | 32
Completed | 29 | 30
Not Completed | 3 | 2
Not completed — Discharged Prior to Study Completion | 2 | 1
Not completed — Participant Opted for Morphine PCA | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the total number of participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.9) | 55 (11.2) | 52.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Average Postoperative Pain Score
Description: Postoperative pain scores were collected once per day during morning rounds for the preceding 24 hours. Participant were asked to provide pain scores for "worst," "average," and "least" pain using the 11-point Numerical Rating Scale (NRS), where 0 represents the absence of pain and 10 is worst possible pain. The average postoperative pain score for each treatment arm is reported.
Time Frame: Participants were followed for the duration of hospital stay, an average of approximately 3 days.
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale | 6.0 (2.2) | 7.3 (2.2)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.0241, Wilcoxon (Mann-Whitney) — A P-value of <0.05 was indicative of statistical significance

2. Secondary Outcome: Worst Postoperative Pain Score
Description: Postoperative pain scores were collected once per day during morning rounds for the preceding 24 hours. Participant were asked to provide pain scores for "worst," "average," and "least" pain using the 11-point Numerical Rating Scale (NRS), where 0 represents the absence of pain and 10 is worst possible pain. The average worst postoperative pain score for each treatment arm is reported.
Time Frame: Participants were followed for the duration of hospital stay, an average of approximately 3 days.
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale | 8.7 (2.0) | 9.0 (1.9)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.4102, Wilcoxon (Mann-Whitney) — A P-value of <0.05 was indicative of statistical significance

3. Secondary Outcome: Least Postoperative Pain Score
Description: Postoperative pain scores were collected once per day during morning rounds for the preceding 24 hours. Participant were asked to provide pain scores for "worst," "average," and "least" pain using the 11-point Numerical Rating Scale (NRS), where 0 represents the absence of pain and 10 is worst possible pain. The average least postoperative pain score for each treatment arm is reported.
Time Frame: Participants were followed for the duration of hospital stay, an average of approximately 3 days.
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale | 4.4 (3.1) | 5.6 (3.0)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.1085, Wilcoxon (Mann-Whitney) — A P-value of <0.05 was indicative of statistical significance

4. Secondary Outcome: 24-Hour Postoperative Opioid Use
Description: Opioid use is defined as the total milligrams of hydromorphone plus other home or oral opioid used per 24 hours, converted to oral morphine equivalents.
Time Frame: For 24 hours following surgery
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: oral morphine mg equivalents
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 29 | 30
oral morphine mg equivalents | 726 (489) | 770 (560)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.7480, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Treatment Related Adverse Events (AEs)
Description: Participants were asked to complete a "Side Effects Checklist" to assess for any unwanted side effects (AEs) of drugs that were administered. The determination of whether or not an AE was treatment related was at the discretion of the Investigator.
Time Frame: Participants were followed for the duration of hospital stay, an average of approximately 3 days.
Population: All randomized participants who completed the study and also completed the Side Effects Checklist.
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 27 | 28
participants
  Respiratory depression | 0 | 0
  Hallucination | 1 | 0
  Pruritis | 5 | 2
  Sedation | 25 | 24
  Nausea | 7 | 5

ADVERSE EVENTS:
Description: Adverse events are reported for all randomized participants who completed the study and also completed the Side Effects Checklist.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/28
Other Adverse Events (participants affected / at risk) | 5/27 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=27) | Placebo (N=28)
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=27) | Placebo (N=28)
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes